CLINICAL TRIAL: NCT06518720
Title: Treatment With Psilocybin for Chronic Neuropathic Pain and Depression (TRANSCEND): An Open-Label Clinical Trial
Brief Title: Treatment With Psilocybin for Chronic Neuropathic Pain and Depression (TRANSCEND)
Acronym: TRANSCEND
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Ishrat Husain, Senior Scientist, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 179-2023
Record Dates: First submitted 2024-07-16; First posted 2024-07-24 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Treatment Resistant Depression; Chronic Pain
Keywords: Psilocybin; Psychedelics; Clinical Trial; Chronic Pain; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Chronic Pain | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psilocybin (25 mg) (Experimental): One capsule of psilocybin 25 mg will be taken orally with a glass of water.
  Interventions: Drug: Psilocybin 25 mg

INTERVENTIONS:
Drug: Psilocybin 25 mg — The psilocybin used in this study meets quality specifications suitable for human research use. The active drug is encapsulated using a hydroxypropyl methylcellulose (HPMC) capsule and contains 25 mg of psilocybin. The psilocybin will be administered once during the trial in combination with supportive therapy.
  Other Names: PEX010

SUMMARY:
Psilocybin, the chemical component of "magic mushrooms", has been administered with psychotherapy in several randomized clinical trials (RCTs) showing large and sustained antidepressant effects.

The purpose of this study is to assess the feasibility, tolerability, and preliminary efficacy of psilocybin therapy for adults with chronic neuropathic pain and co-morbid treatment resistant depression.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 65 years old;
2. Are outpatients;
3. Must be deemed to have capacity to provide informed consent;
4. Must sign and date the informed consent form;
5. Stated willingness to comply with all study procedures;
6. Ability to read and communicate in English, such that their literacy and comprehension is sufficient for understanding the consent form and study questionnaires, as evaluated by study staff obtaining consent;
7. Primary DSM-5 diagnosis of non-psychotic MDD, single or recurrent, based on the Structured Clinical Interview for DSM-5 (SCID-5) administered at the first screening visit;
8. Participants diagnosed with treatment-resistant depression defined as individuals with a baseline HamD-17 score > 14 and that have not responded to two or more separate trials of antidepressants at an adequate dosage and duration (an antidepressant resistance rating score of three or more is considered an adequate trial) based on the Antidepressant Treatment History Form (ATHF) (Sackeim & Sackeim, 2001); there is no upper limit on the number of treatment failures;
9. Diagnosis of chronic neuropathic pain as determined by a pain specialist and confirmed with the standardized Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) questionnaire25
10. Moderate-to-severe neuropathic pain determined by Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference score of > 6026, as well as mean pain intensity scores > 5 on a numeric rating scale27
11. Previous trials of at least two medications recommended in the Canadian consensus guidelines on the management of neuropathic pain with no self-reported meaningful improvement in symptoms
12. Ability to take oral medication;
13. Individuals with an eGFR above 40mL/min/1.73m2 and all blood work on clinical laboratory tests assessed as not clinically significant by study delegate physician at Screening (V1)
14. Individuals who are capable of becoming pregnant: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation;
15. Individuals who are willing to taper off current antidepressant and antipsychotic medications for a minimum of 2-weeks (or more depending on the medication) prior to Baseline (V2) and for the duration of the study and whose physician confirms that it is safe for them to do so; and
16. Agreement to adhere to Lifestyle Considerations (section 4.5) throughout study duration.

Exclusion Criteria:

1. Pregnant as assessed by a urine pregnancy test at Screening (V1) or individual's that intend to become pregnant during the study or are breastfeeding;
2. Treatment with another investigational drug or other intervention within 30 days of Screening (V1);
3. Have initiated psychotherapy in the preceding 12 weeks prior to Screening (V1);
4. Have a DSM-5 diagnosis of substance use disorder (recreational use of tobacco, alcohol, cannabis and prescribed opioids are permitted) within the preceding 6 months;
5. Have active suicidal ideation with intent and plan as determined by item 3 of the HamD-17;
6. Any DSM-5 lifetime diagnosis of a schizophrenia-spectrum disorder; obsessive-compulsive disorder, psychotic disorder (unless substance induced or due to a medical condition), bipolar I or II disorder, paranoid personality disorder, borderline personality disorder, or neurocognitive disorder as determined by medical history and the SCID-5 clinical interview;
7. Any first-degree relative with a diagnosis of schizophrenia-spectrum disorder; psychotic disorder (unless substance-induced or due to a medical condition); or bipolar I or II disorder as determined by the family medical history form and discussions with the participant;
8. Presence of a relative or absolute contraindication to psilocybin, including a drug allergy, recent stroke history, uncontrolled hypertension, low or labile blood pressure, recent myocardial infarction, cardiac arrhythmic, severe coronary artery disease, or moderate to severe renal or hepatic impairment.
9. Presence of baseline prolonged QTc or Torsade de Pointes as measured by the ECG or a history of long QTc syndrome or related risk factors;
10. Individuals who are currently taking methadone, buprenorphine or > 100 milligrams of morphine (or morphine equivalents).
11. Any other clinically significant physical illness including chronic infectious diseases or any other major concurrent illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if they take part in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants recruited, enrolled and retained (feasibility) and the number of serious adverse events and serious adverse drug reactions associated with administration of 25 mg of psilocybin (safety). | 24 Months
  Percentage of participants recruited, enrolled and retained over 24 months. Number of serious adverse events and serious adverse drug reactions associated with psilocybin 25 mg.

SECONDARY OUTCOMES:
Change in the Montgomery-Åsberg Depression Rating Scale (MADRS) from Baseline to 1-week post-treatment. | Baseline (Visit 2, Day 0) to 1-week post-treatment (Visit 4, Day 7).
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinician-rated scale that measures depression severity. This measure has 10 items rated from 0-6. The lowest possible score is 0 and highest possible score is 60. Higher composite scores represent a more severe condition/ worse outcomes.

OTHER OUTCOMES:
Change in Patient Reported Outcomes Measurement Information System-Pain Intensity Scale (PROMIS-PI) from Baseline to 1-week post-treatment. | Baseline (Visit 2, Day 0) to 1-week post-treatment (Visit 4, Day 7).
  The Patient Reported Outcomes Measurement Information System-Pain Intensity Scale (PROMIS-PI) is a participant-rated scale that measures intensity of pain experienced by the participant in the past seven days. Presented on a visual analogue scale of 0-10, scores range from 0= no pain to 10=worst imaginable pain. A score of 5 or greater indicates moderate to severe pain intensity.
Change in Patient Reported Outcomes Measurement Information System- Pain Interference Scale (PROMIS-Interference) from Baseline to 1-week post-treatment. | Baseline (Visit 2, Day 0) to 1-week post-treatment (Visit 4, Day 7).
  The Patient Reported Outcomes Measurement Information System- Pain Interference Scale (PROMIS-Interference) is a participant rated scale that aims to identify how much an individual's physical pain has interfered with emotional, social and cognitive domains of living. A T-Score greater than 50 indicates higher pain interference than the general population.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Ishrat Husain, MBBS, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT06518720/Prot_SAP_000.pdf